CLINICAL TRIAL: NCT05891223
Title: The Effect of "Mindfulness-Based Compassionate Life Training" for University Students Affected by the Earthquake on Coping With Earthquake Trauma Stress and Grief Process
Brief Title: The Effect of "Mindfulness-Based Compassionate Life Training" for University Students Affected by the Earthquake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Suheyla YARALI, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: suheylayaralı
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Earthquake; Trauma; Stress, Psychological
Keywords: Mindfulness; self-compassion; Trauma; Psychological
MeSH Terms: conditions — Wounds and Injuries; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Session 1: How We Evolved - Threat, Impulse, and Soothing Systems (Experimental): * A "breath break with kindness" is practiced.
  * Encourage them to think about how threat, impulse and sedative systems have developed in their own lives.
  * A "safe place" application is made.
  * "Courtesy meditation" is done.
  Interventions: Other: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
- Session 2: Threat and Self-Compassion (Experimental): * A "breath break with kindness" is practiced.
  * "Building a compassionate relationship with resilience" and "kindness meditation: a benevolent" practices are made.
  * "A hand on your heart" and "a compassionate comrade" practices are made.
  Interventions: Other: Session 2: Threat and Self-Compassion
- Session 3: Unraveling the Knots of Desire and Patterns Agenda (Experimental): * Talk about homework.
  * A "breath break with kindness" is practiced.
  * "Establishing a compassionate relationship with desire", "guided meditation to discover the inner pattern", "courtesy meditation: a good friend" practices are made.
  Interventions: Other: Session 3: Unraveling the Knots of Desire and Patterns
- Session 4: Internalizing compassion (Experimental): * "Pretend-to-pretend" practice is made for participants to observe themselves.
  * In addition to the previous practices, the practice of "internalizing compassion" is made in order to increase their expanded mindfulness.
  * "Courtesy meditation: a neutral person", "kindness towards your body", which is based on mindfulness practices and increases body awareness and mindful movement, is carried out. During the day, they will be informed that they should do the "walking with kindness" practice on their own.
  Interventions: Other: Session 4: Internalizing compassion
- Session 5: Me and others - Expanding the circle (Experimental): * A "compassionate letter" application is made by asking participants to think about a situation they encountered recently or some time ago and is still causing distress. It is explained that they can gain insight with this application.
  * "Courtesy meditation: the 'difficult' person", "compassion and breathing: yourself" and "compassionate breathing: others" practices are made.
  Interventions: Other: Session 5: Me and others - Expanding the circle
- Session 6: Growing happiness (Experimental): * "Revisiting the good" practice is carried out to define the five sense organs for the participants.
  * "Forgiveness", "Asking for forgiveness", "forgiving others", "gratitude" practices are carried out.
  * The practice is expanded as "kindness meditation: groups and all beings".
  Interventions: Other: Session 6: Growing happiness
- Session 7: Weaving Wisdom and Compassion into Daily Life (Experimental): * Participants are made to choose a day in their life and allow a few minutes to pause in a mindful way.
  * "A breather for wise and compassionate action", "calmness meditation" and "joy sharing meditation" practices are carried out.
  Interventions: Other: Session 7: Weaving Wisdom and Compassion into Daily Life
- Session 8: Living with the Heart (Experimental): * The participants are told about the applications that they can apply for, where they need help to develop compassion towards self-healing skills, and the whole training is evaluated.
  * The "river of life" application, which evaluates mindfulness in depth, is carried out.
  * An overall summary of the 8-session study is made and feedback is received.
  Interventions: Other: Session 8: Living with the Heart

INTERVENTIONS:
Other: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems — The practice of "Breath break with kindness" will be applied for 5 minutes. Afterwards, 15 minutes of information on threats, impulses and soothing systems, "A safe place" application for 11 minutes, "Courtesy meditation" for 10 minutes. After each application, 10 minutes of feedback will be received from the participants.
  Arms: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
Other: Session 2: Threat and Self-Compassion — The practice of "breathing with kindness" will be done for 7 minutes. The practice of "Building a compassionate relationship with resilience" will be held for 12 minutes, and the practice of "Kindness meditation: a benevolent" will take place for 11 minutes. "A hand over your heart" application will be made for 3 minutes and "A compassionate comrade" application will be done for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 2: Threat and Self-Compassion
Other: Session 3: Unraveling the Knots of Desire and Patterns — The practice of "breathing with kindness" will be done for 7 minutes. "Building a compassionate relationship with desire" 12 minutes, "Guided meditation to discover the inner pattern" 10 minutes and "Courtesy meditation: a good friend" 11 minutes. Except for the "breath break with kindness" application, 3 minutes of feedback will be received from the participants after each application.
  Arms: Session 3: Unraveling the Knots of Desire and Patterns Agenda
Other: Session 4: Internalizing compassion — The "pretend-to-be" practice for the participants to observe themselves will be made for 10 minutes. The practice of "internalizing compassion" will be done for 7 minutes, "kindness meditation: a neutral person" practice for 10 minutes, and "kindness towards your body" for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 4: Internalizing compassion
Other: Session 5: Me and others - Expanding the circle — The "a compassionate letter" practice with the participants will continue for 15 minutes. "Courtesy meditation: the 'difficult' person" 8 minutes, "compassion and breathing: yourself" 10 minutes and "compassionate breathing: others" 7 minutes. A "compassionate break" application is performed for 7 minutes.
  Arms: Session 5: Me and others - Expanding the circle
Other: Session 6: Growing happiness — The practice of "Revisiting the good" is carried out for 10 minutes with the participants. "Forgive yourself", "wish for forgiveness", "forgive others", "gratitude" practices will be held for 5 minutes each and will take 20 minutes in total. "Courtesy meditation: groups and all beings" will be practiced for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 6: Growing happiness
Other: Session 7: Weaving Wisdom and Compassion into Daily Life — Participants will be given 10 minutes to choose a day in their life and allow a few minutes to pause mindfully. The practice of "a breather for wise and compassionate action" is 10 minutes, the practice of "calmness meditation" is 8 minutes, and the practice of "sharing the joy meditation" is 8 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 7: Weaving Wisdom and Compassion into Daily Life
Other: Session 8: Living with the Heart — The participants are told about the applications they can apply for, where they need help to develop compassion towards self-healing skills, and the entire training will be evaluated for 20 minutes. The "river of life" application is carried out for 20 minutes. 10 minutes of feedback will be received after the application.
  Arms: Session 8: Living with the Heart

SUMMARY:
In this study, aimed to determine the effect of "Mindfulness Based Compassionate Life Training" given to university students on coping with post-earthquake trauma stress and grief process. According to the experimental design with pre-test and post-test control group, the participants selected from the universe will be assigned to the experimental and control groups impartially. In this study, a priori power analysis will be performed to determine the sample size. For the independent groups, in which the effect of "Mindfulness-Based Compassionate Life Training" on coping with post-earthquake trauma stress and grief will be compared, 80% power will be achieved at a significance level of 0.05 at a 95% confidence interval. A total of 68 participants will be reached by taking into account data losses and including 30% backup sample in the research. Participants included in the study will be numbered from 1 to 68 and 34 experimental and 34 control groups will be created from www.random.org.

Pre-test data will be collected before applying to earthquake survivors in the experimental group and control group. 8 sessions of Mindfulness Based Compassionate Life training will be given to earthquake survivors in the experimental group. Training sessions will be held online. For its effectiveness and continuity, each session will be held between 3 days and 7 days. One week after the Mindfulness-Based Compassionate Living training (after 8 sessions were completed), the "Post-earthquake Trauma Stress Level Determination Scale (NSSTDBÖ)", "The Grief Scale" was administered to the earthquake survivors. The "Self-Compassion Scale Short Form (STS-F)" post-test will be filled in by face-to-face interview. Post-test data from the experimental and control groups will be obtained simultaneously.

DETAILED DESCRIPTION:
Research data will be collected face to face by researchers. 68 earthquake survivors who meet the inclusion criteria (to be studying at a university, to be affected by the earthquake, to be willing to participate in the study, to be open to communication and cooperation) will be included in the study. The descriptive features form consisting of 8 questions for data collection, "Post-earthquake Trauma Stress Level Detection Scale", "Mourning Scale". "Self-Compassion Scale Short Form (STS-F)" will be used. Research data will be collected as a pre-test and post-test for 1 month. Those who do not regularly participate in the Mindfulness-Based Compassionate Living training will be excluded from the study. The research will be carried out with 68 participants, 34 in the experimental group and 34 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Having a university nursing education
* Being affected by the earthquake
* Willingness to participate in the study
* Being open to communication and cooperation

Exclusion Criteria:

* Not attending sessions regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-06-05 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | [Time Frame: up to 1 day]
  The form consists of 8 questions containing information about the students affected by the earthquake created by the researcher within the scope of the literature. The form created, gender, place of residence, the state of being together with the parents, whether the parents are alive or not, the place where they stayed during the earthquake (home, dormitory, etc.) to what extent they were affected by the earthquake, the status of losing a relative in the earthquake, the status of receiving psychological support after the earthquake, more It includes questions about experiencing a traumatic event before and having a previously diagnosed psychiatric illness.

SECONDARY OUTCOMES:
Post-earthquake Trauma Stress Level Scale (DSSTDBÖ) | [Time Frame: up to 5 week ]
  DSTDBÖ is a tool developed by Tanhan and Kayri (2013) to measure the stress levels experienced by individuals after an earthquake. The scale consists of 20 items. The scale was arranged with a 5-point Likert-type rating of "strongly disagree", "little agree", "moderately agree", "strongly agree".
  and "totally agree" format. The lowest score that can be obtained from the scale is 20 and the highest score is 100. The increase in the scores obtained from the scale shows that the individuals' level of being affected by the earthquake also increases. The internal consistency coefficient (Cronbach's alpha) of the DSDTDS was found to be .87.

OTHER OUTCOMES:
Grief Scale | [Time Frame: up to 5 week ]
  The grief scale developed by Balcı (2006) measures the physical, emotional, intellectual and behavioral changes that occur in the individual after the loss of a loved one or persons. The scale consists of 35 items and four sub-dimensions. Items 11, 13 and 17 are reverse coded. Individuals are given statements about the situations they may experience in the face of a separation or loss, on a scale of 1-5, (5) Always, (4) Often, (3) Occasionally, (2) Rarely, (1) They are asked to rank as Never. The highest score that can be obtained from the entire scale is 175, and the lowest score is 35. The scale has no cut-off point. It is stated that the higher the score, the higher the level of grief. The Cronbach Alpha internal consistency coefficient for the internal consistency reliability of the scale is .96.
Short Form of Self-Compassion Scale (SSS-C) | [Time Frame: up to 5 week ]
  The Turkish validity and reliability of the scale developed by Neff (2003) was made by Yıldırım and Sarı in 2018. The scale was confirmed to have a structure consisting of 11 items, a single dimension, and two complementary components (positive component and negative component). The internal consistency coefficient of the scale was calculated as .75. SSS-F Total score is used to measure self-compassion. It is stated that as the score increases, the level of Self-compassion increases. This scale was used by Liu et al. was used as a measurement tool in the evaluation of individuals who experienced earthquakes. (Liu., et all, 2021)